CLINICAL TRIAL: NCT02976207
Title: Long Follow up on Patients With Obstructive Sleep Apnea That Undergo Diagnosis and Surgical Treatment
Acronym: OSA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 55-2015
Record Dates: First submitted 2016-11-08; First posted 2016-11-29 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: OSA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years

GROUPS / COHORTS (1):
- OSA diagnosed patients: patients at the age range of 18-90, male or female, who are diagnosed as suffering from OSA and are surgery candidates for their condition.

SUMMARY:
Long follow up on patients with obstructive sleep apnea that undergo diagnosis and surgical treatment

DETAILED DESCRIPTION:
Drug induced sleep endoscopy (DISE) is increasingly performed procedure, offering dynamic upper airway evaluation during artificial sleep before surgical treatment for patients with obstructed

.)OSA(sleep apnea

* Aim: To evaluate the value of DISE for tailoring the proper treatment for patients with snoring and OSA DISE is a safe procedure, easily practicable, valid and reliable. We consider it a fundamental clinical procedure that is essential before choosing the surgical treatment. Our results so far suggest that a multilevel collapse is significantly associated with higher apnea hypopnea index values. We think that the weight did not play a significant role in RDI (Respiratory Disturbance Index) reduction. Our results till now show tailored surgery based on DISE may leverage sleep surgeries outcome significantly presenting 70% success rate based
* on our experience We therefore want to evaluate the patients in a long follow up period

ELIGIBILITY:
Inclusion Criteria:

* Fully diagnosed patients with OSA.
* Patients who are candidates for a surgery as a treatment to their condition.

Exclusion Criteria:

* Pregnancy
* Patients who are not OSA surgery candidates.
* Patients with high surgical risk.
* Patients with hematological or oncological background.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients at the age range of 18-90, male or female, who are diagnosed as suffering from OSA and are surgery candidates for their condition.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-01; Primary Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of daytime sleepiness- using Epworth sleepiness scale questionnaire | up to 3 years after surgery
Sleep quality assessment questionnaire | up to 3 years after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yafe medical center, Hadera, Hadera, Israel